CLINICAL TRIAL: NCT00201721
Title: Phase II Trial of Pentostatin, and Rituximab With and Without Cyclophosphamide for Previously Untreated B-Chronic Lymphocytic Leukemia (CLL)
Brief Title: Pentostatin, and Rituximab With and Without Cyclophosphamide for Previously Untreated B-Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: Astex Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, John Byrd, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-0143; NCT00423423 (obsolete NCT alias)
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: B-Chronic Lymphocytic Leukemia
Keywords: Previously Untreated
MeSH Terms: conditions — Leukemia, B-Cell | interventions — Pentostatin; Rituximab; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Pentostatin — 2 mg/m2 IV over 30 minutes in 250 mL NS on day 1 during cycles 1-6.
  Other Names: Nipent®
Drug: Rituximab — For the first week only: Day 1 of therapy 100 mg IV over 4 hours. Day 3 of therapy 375 mg/m2 IV at 50 mg/hr and increase by 100 mg/hr at 30-minute intervals to a maximum of 400 mg/hr. Day 5 of therapy 375 mg/m2 IV at 100 mg/hr for the first 15 minutes the remainder goes in at 45 minutes. The remaining weeks 375 mg/m2 will be repeated as a single IV infusion Day 1 of Week 4, 7, 10, 13 and 16 during cycles 2-6.
  Other Names: RITUXAN®
Drug: Cyclophosphamide — 600 mg/m2 IV in 250 mL NS over 30 minutes on day 1 cycles 1-6
  Other Names: CTX

SUMMARY:
This study aims to assess the rate of complete and overall response using rituximab and pentostatin with and without cyclophosphamide, to monitor and assess toxicity of this regimen, and to determine the overall and progression-free survival in CLL patients

DETAILED DESCRIPTION:
Rationale: Research indicates that both cyclophosphamide and pentostatin work synergistically against cancer cells and have a high response rate against chronic lymphocytic leukemia (CLL) without creating severe side effects in patients. In addition, studies have shown that rituximab, a therapy that targets the immune system, has the highest efficacy against CLL and the lowest toxicity rate when compared with other immunotherapy drugs. Studies also show that rituximab enhances the efficacy of the chemotherapy agents cyclophosphamide and pentostatin. This study offers the combination of immunotherapy with two promising chemotherapy agents against CLL.

Purpose: This study is evaluating the efficacy and safety of combination treatment with cyclophosphamide, pentostatin, and rituximab in patients with CLL. Several tests evaluating the genetic and molecular components of CLL will also be performed. Some of these tests will be conducted before, during, and after treatments to assess changes resulting from the study drugs. Each patient's outcome will be assessed in relation to various aspects of their genes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of B-CLL (no mantle cell)
* Must have active disease
* Age >=18 yo
* ECOG 0-3
* No radiation or surgery <4 weeks

Exclusion Criteria:

* Any of the following comorbid conditions:

  * New York Heart Association Class III or IV heart disease
  * Recent myocardial infarction (<1 month)
  * Uncontrolled infection
  * Active infection with the human immunodeficiency virus (HIV/AIDS) as further severe immunosuppression with this regimen may occur.
* Pregnant or nursing women
* Men or women of child bearing potential must use adequate contraception.
* Active primary malignancy requiring treatment or limits survival to ≤2 years.
* Any radiation therapy ≤4 weeks prior to study entry.
* Any major surgery ≤4 weeks prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2002-07; Primary Completion 2006-07 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
To assess the rate of complete and overall response using rituximab and pentostatin with and without cyclophosphamide. | up to 5 years
  For this evaluation, patients will be classified as complete responders if either of the following types of response are documented
  * CCR (Clinically based complete remission) denotes NED (No Evidence of Disease) based on baseline clinical parameters.
  * CR denotes CCR and, in bone marrow, no nodules and <30% lymphocytes.

SECONDARY OUTCOMES:
To monitor and assess toxicity of this regimen. | up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: John Byrd, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University, Columbus, Ohio, United States

REFERENCES:
- [Background] Kay NE, Geyer SM, Call TG, Shanafelt TD, Zent CS, Jelinek DF, Tschumper R, Bone ND, Dewald GW, Lin TS, Heerema NA, Smith L, Grever MR, Byrd JC. Combination chemoimmunotherapy with pentostatin, cyclophosphamide, and rituximab shows significant clinical activity with low accompanying toxicity in previously untreated B chronic lymphocytic leukemia. Blood. 2007 Jan 15;109(2):405-11. doi: 10.1182/blood-2006-07-033274. Epub 2006 Sep 28. PMID 17008537
- [Result] Kay NE, Wu W, Kabat B, LaPlant B, Lin TS, Byrd JC, Jelinek DF, Grever MR, Zent CS, Call TG, Shanafelt TD. Pentostatin and rituximab therapy for previously untreated patients with B-cell chronic lymphocytic leukemia. Cancer. 2010 May 1;116(9):2180-7. doi: 10.1002/cncr.25028. PMID 20187101
- [Result] Shanafelt TD, Lin T, Geyer SM, Zent CS, Leung N, Kabat B, Bowen D, Grever MR, Byrd JC, Kay NE. Pentostatin, cyclophosphamide, and rituximab regimen in older patients with chronic lymphocytic leukemia. Cancer. 2007 Jun 1;109(11):2291-8. doi: 10.1002/cncr.22662. PMID 17514743
- See also: Jamesline — http://cancer.osu.edu